CLINICAL TRIAL: NCT01980238
Title: Defunctioning Cannula Ileostomy After Lower Anterior Resection of Rectal Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hua hanju, Doctor, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cannula ileostomy
Record Dates: First submitted 2013-10-23; First posted 2013-11-08 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Rectal Neoplasms
Keywords: LAR; anastomotic leakage; Cannula ileostomy; loop ileostomy
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak | interventions — Ileostomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- cannula ileostomy (Experimental): After LAR, experimental group will accept cannula ileostomy. Operation has described in the Detailed Description.
  Interventions: Device: cannula ileostomy; Device: LAR
- loop ileostomy (Active Comparator): After LAR, active comparator group will accept loop ileostomy. This operation is well known by colorectal surgeons.
  Interventions: Device: loop ileostomy; Device: LAR

INTERVENTIONS:
Device: cannula ileostomy
  Arms: cannula ileostomy
Device: loop ileostomy
  Arms: loop ileostomy
Device: LAR
  Other Names: Low anterior resection

SUMMARY:
Most surgeons suggest the use of fecal diverting to address the high morbidity and mortality associated with anastomotic leakage (AL) in patients with high risk factors on AL who are undergoing anterior resections. Although debate about the use of defunctioning stoma continues, meta-analyses and randomized multicenter trial results support the use of defunctioning stoma in lower anterior resection(LAR). This exploratory study was conducted to evaluate the efficacy and safety of a new diversion method called spontaneously closed cannula ileostomy (SCCI), which was designed to protect rectal anastomosis in patients with high risk factors on AL. Results of SCCI were compared to those of the loop ileostomy (LI) method.

DETAILED DESCRIPTION:
After low anterior resection(LAR), in the LI group, the operation method was done as surgeons all known. In the cannula ileostomy group, a double row of concentric purse-string sutures were placed in the ileum wall using 3-0 absorbable suture. The diameters of the purse-string rings were about 10 mm and 20 mm, respectively. The investigators then made a small incision within the inner purse-string and inserted the trachea cannula into the proximal end of the ileum. The inner purse-string suture then was tied, followed by the outer purse-string suture. The outer purse string should capsulate the inner purse string to prevent leakage. Normal saline was injected into the air bag until the ileum wall began to turn pale. The investigators then pulled the cannula out through the abdominal wall. The incision site in the ileum was approximated to the inner abdominal wall and extraperitonized by fixing the mobilized ileum wall around the cannula to the inner abdominal wall. This was accomplished using 3-4 interrupted sutures.

In the LI group, patients accepted reversal operation at least 3 months after operation if operation condition permission.

In the cannula ileostomy group, the cannula will be removed after 3-4 weeks. If anastomotic leakage occurred, The investigators will keep the cannula until the anastomotic leakage was cured.

ELIGIBILITY:
Inclusion Criteria:

1. Rectal Tumor After Low Anterior Resection the Anastomosis Located extraperitoneal.
2. Intraperitoneal Anastomosis Who Used of Glucocorticoid or Accepted Neoadjuvant Chemoradiotherapy.
3. Patients Agreed to Undergo the Canula Ileostomy or Loop Ileostomy Procedure

Exclusion Criteria:

1. Bowel Preparation is Satisfied Before Operation(This Means That if Surgeons Find That There is Much Feces Left in the Colon,the Patient Will be Excluded)
2. positive air leakage test
3. fractured anastomotic rings

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
anastomotic leakage, reoperation and mortality rate | about in 3 months after operaion.
  Anastomotic leakage(AL) is the main complication after LAR.AL is defined as a defect of intestinal wall integrity at the colorectal or coloanal anastomotic site (including suture and staple lines of the neorectal reservoirs) leading to communication between intra- and extraluminal compartments. When AL occurred, whether this patient need reoperation is determined by the clinical manifestation. Reoperation rate and mortality are two key index to evaluate the effect and safety of cannula ileostomy.

SECONDARY OUTCOMES:
ileus rate | during the follow time(about 6 months after operaion)
  Another main operation complication was intestinal obstruction. Ileus conclude two types: temporally ileus and intractable ileus. Temporally ileus can be treated by conservative treatment and intractable ileus need reoperation.Ileus usually is caused by intestinal adhesion. But in cannula ileostomy group, ileus maybe caused by the cannula obstruction.

OTHER OUTCOMES:
hospital stays and costs | from admission time to discharge time(about 7-14days)
  In loop ileostomy group, hospital stays and costs include the readmission to close the stoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Colorectal Surgery, First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China